CLINICAL TRIAL: NCT03409822
Title: The Effectiveness of Intraoperative Non-invasive Hemoglobin Monitoring in Parturients With Placenta Previa Undergoing Cesarean Section: Prospective Observational Study
Brief Title: Non-invasive Hemoglobin Monitoring in Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Principle investigator, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hb Csec
Record Dates: First submitted 2018-01-09; First posted 2018-01-24 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Placenta previa (Other)
  Interventions: Device: Masimo SpHb™ monitor

INTERVENTIONS:
Device: Masimo SpHb™ monitor — Attach the Masimo Rainbow SET® Radical-7 ™ pulse oximeter probe to the third or fourth finger and perform a Masimo SpHb ™ monitor.

SUMMARY:
Non-invasive hemoglobin monitoring will be performed in patients who underwent cesarean section with placenta previa and this will be compared with actual laboratory findings.

The investigators will investigate whether noninvasive hemoglobin monitoring can adequately reflect the massive bleeding that occurs within a short period of time and find out if it matches the actual laboratory findings.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Elective Cesarean section
* Placenta previa

Exclusion Criteria:

* Decline of consent
* Peripheral vascular disease
* Cyanosis due to congenital heart disease
* Refusal of transfusion
* Mental retardation

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
The change of total hemoglobin | 10 min before operation, 10 min after operation, 1 min after skin incision, 1 min after delivery of baby, 1 min after removal of placenta, 1 min after skin closure

SECONDARY OUTCOMES:
The change of oxygen content | 10 min before operation, 10 min after operation, 1 min after skin incision, 1 min after delivery of baby, 1 min after removal of placenta, 1 min after skin closure
The change of methemoglobin | 10 min before operation, 10 min after operation, 1 min after skin incision, 1 min after delivery of baby, 1 min after removal of placenta, 1 min after skin closure
The change of carboxyhemoglobin | 10 min before operation, 10 min after operation, 1 min after skin incision, 1 min after delivery of baby, 1 min after removal of placenta, 1 min after skin closure
The change of pleth variability index | 10 min before operation, 10 min after operation, 1 min after skin incision, 1 min after delivery of baby, 1 min after removal of placenta, 1 min after skin closure
The change of perfusion index | 10 min before operation, 10 min after operation, 1 min after skin incision, 1 min after delivery of baby, 1 min after removal of placenta, 1 min after skin closure

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univ. Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea